CLINICAL TRIAL: NCT06851039
Title: Effects of the Resistant Starch and Sodium Butyrate Supplementation on the Respiratory and Cardiovascular Autonomic Control in Humans
Brief Title: Effects of the Short-Chain Fatty Acids-Targeted Dietary Interventions on the Selected Autonomic Functions in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Rafał Seredyński, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STM.A090.20.110
Record Dates: First submitted 2025-02-13; First posted 2025-02-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: resistant starch; short-chain fatty acids; gut microbiota; peripheral chemoreflex; arterial baroreflex; autonomic nervous system

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- potato starch (Experimental)
  Interventions: Dietary Supplement: Potato starch supplementation
- sodium butyrate (Experimental)
  Interventions: Dietary Supplement: Sodium butyrate supplementation
- accessible maze starch (Placebo Comparator)
  Interventions: Dietary Supplement: Accessible starch supplementation

INTERVENTIONS:
Dietary Supplement: Potato starch supplementation — Participants will receive potato starch supplement, undergoing gut microbial fermentation and acting as an endogenous source of the short-chain fatty acids, including butyrate. Effects of these compounds on the selected autonomic functions (i.e. cardio-respiratory control) will be further investigated.
  Arms: potato starch
Dietary Supplement: Sodium butyrate supplementation — Participants will receive sodium butyrate supplement, acting as an exogenous source of the short-chain fatty acid butyrate. Effects of such compound on the selected autonomic functions (i.e. cardio-respiratory control) will be further investigated.
  Arms: sodium butyrate
Dietary Supplement: Accessible starch supplementation — Participants will receive the accessible (digestible) waxy maze starch as placebo.
  Arms: accessible maze starch

SUMMARY:
Recent data feature short-chain fatty acids (SCFAs), products of gut microbial fermentation, as modulators of the blood pressure of the host. Such modulation may evoke (or arise from) changes in the autonomic reflexive mechanisms, but the link remains unexplored. Therefore, the study aims to explore potential relationship between the dietary intervention-induced changes in the SCFA plasma/fecal content and alterations in the sensitivity of the cardio-respiratory autonomic reflexes.

In this cross-over, placebo-controlled study, a group of healthy volunteers will undergo three distinct stages of a four-week dietary intervention, separated by at least two weeks of washout periods. During each stage, participants will receive one of the following interventions:

* raw potato starch (a source of resistant type 2 starch, which is a substrate for the endogenous production of SCFAs)
* sodium butyrate (a direct, exogenous source of this SCFA)
* an amylase-accessible waxy maze starch (a placebo). Plasma and fecal SCFA concentrations will be measured, along with the comprehensive evaluation of the cardio-respiratory parameters and the sensitivity of the autonomic reflexive mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years

Exclusion Criteria:

* chronic disease of the nervous, cardiovascular or respiratory system
* disease of the digestive system, including history of the intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance and other malabsorption disorders
* blood pressure-lowering treatment within the past year
* tobacco smoking within the past year
* antibiotic/probiotic treatment and laxative/prokinetic usage in three months preceding the anticipated enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Arterial baroreflex sensitivity | From the beginning to the end of a supplementation period at 4 weeks.
  Arterial baroreflex sensitivity, measured with a neck chamber technique.
Peripheral chemoreflex sensitivity | From the beginning to the end of a supplementation period at 4 weeks.
  Peripheral chemoreflex sensitivity, measured with the transient hypoxia test.

SECONDARY OUTCOMES:
Plasma short-chain fatty acids | From the beginning to the end of a supplementation period at 4 weeks.
  Plasma level of short-chain fatty acids, evaluated with high-performance liquid chromatography.

CONTACTS AND LOCATIONS:
Locations (1):
- Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
This is a small trial which includes solely healthy volunteers. Therefore, data will not be shared at this instance.